CLINICAL TRIAL: NCT05176847
Title: Increasing Social Support for Weight Loss Through the Use of Social Gaming and Points: The Mobile Intervention for Food and Exercise (mLIFE) Study
Brief Title: The Mobile Lifestyle Intervention for Food and Exercise Study
Acronym: mLIFE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Brie Turner-McGrievy, Associate Professor, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Pro00109784; 1R01DK129302 (NIH)
Record Dates: First submitted 2021-12-16; First posted 2022-01-04 (Actual); Results first posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Overweight and Obesity; Type2 Diabetes
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gamified mLIFE app group (Experimental): Participants allocated to this group will be provided with elements of social gaming and healthy competition within the mLIFE app.
  Interventions: Behavioral: Podcasts and tips of the day (within app); Behavioral: mLIFE app (self-regulation features); Behavioral: mLIFE app (social support features)
- standard mLIFE app (Active Comparator): Participants in this group will receive the same intervention as the experimental group, but some features of the App will not facilitate gaming or competition.
  Interventions: Behavioral: Podcasts and tips of the day (within app); Behavioral: mLIFE app (self-regulation features); Behavioral: standard mLIFE app (social support features)

INTERVENTIONS:
Behavioral: Podcasts and tips of the day (within app) — Participants will receive twice weekly podcasts and daily tips of the day, with nutrition and exercise information, audio diary and goal setting.
Behavioral: mLIFE app (self-regulation features) — Diet (track by in app database), physical activity (tracked with FitBit and synced with mLIFE app), and weight (tracked with FitBit scale and synced with mL app) tracking app components. App notifications and reminders and newsfeeds.
Behavioral: mLIFE app (social support features) — The gamified mLIFE app contains several components to help facilitate social gaming and support. This includes a newsfeed, to view the progress of other users, the ability to send others encouragement ("likes/thumbs-up") for achieving goals, user-to-user messaging system so active users of the app will be prompted to select send encouraging messages to other group members.
  For the experimental group, the app also includes features that facilitate healthy competition among participants through receipt of points for provision of social support and tracking health behaviors.
  Arms: Gamified mLIFE app group
Behavioral: standard mLIFE app (social support features) — The standard mLIFE app has the ability to send others encouragement ("likes/thumbs-up") for achieving goals and a user-to-user messaging system so active users of the app will be prompted to select send encouraging messages to other group members.
  Arms: standard mLIFE app

SUMMARY:
The goal of the study is to examine long term sustained weight loss digital intervention in a diverse cohort of adults with overweight/obesity. The intervention includes social gaming (using game-like elements in nongame contexts to promote supportive social interactions and openness to positive behavioral influences) to reward behaviors, such as self-monitoring and social support.

Investigators will accomplish objectives and test hypotheses by following two specific primary aims:

1. Determine if the intervention plus gaming produces significantly more weight loss at 12 months than the same intervention without gaming among 240 adults with overweight or obesity and ≥3 T2DM risk factors.
2. Examine the differences in social support provision and receipt between groups at 12 months.

DETAILED DESCRIPTION:
This is a 1-year behavioral intervention with standardized behavioral content that reinforces self-monitoring behavior delivered via twice-weekly podcasts, tips of the day, weight, physical activity and diet daily tracking. The mLife App will also encourage and facilitate social support among participants (to both groups).

Participants will be randomized to one of two groups: 1) a gamified mLIFE app (n=120) or 2) regular mLIFE app (n=120). Participants will attend a study orientation, complete all baseline measures, be randomized, and then attend a training session for their group. In addition, participants will complete assessment at 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Must be between 18-65 years old
* ≥3 T2DM risk factors (as defined by the American Diabetes Association)
* Own and use a smartphone with a data plan
* BMI must be between 25-49.9 kg/m2
* Must be willing to reduce caloric intake and increase physical activity
* Not currently participating in a weight loss study in a weight loss program
* Be free of major health or psychiatric diseases, drug or alcohol dependency.
* No current use of medications that may impact blood glucose

Exclusion Criteria:

* Over the age of 65 years old
* Currently participating in a weight loss program
* Has lost more than 10 pounds in the past 6 months
* Diagnosed with type 2 diabetes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-07-12 (Actual); Study Completion 2025-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brie Turner-Mcgrievy, Principal Investigator — University of South Carolina
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Turner-McGrievy G, Monroe C, Delgado-Diaz C, Aydin HZ, DuBois K, Kim Y, Valafar H, Wilcox S. Incentivizing social support in the randomized mobile Lifestyle Intervention for Food and Exercise study: the impact of gamification on social support perceptions, provision, and receipt. Transl Behav Med. 2026 Jan 7;16(1):ibaf086. doi: 10.1093/tbm/ibaf086. PMID 41498406
- [Derived] DuBois KE, Delgado-Diaz DC, McGrievy M, Valafar H, Monroe C, Wilcox S, Turner-McGrievy G. The Mobile lifestyle intervention for food and exercise (mLife) study: Protocol of a remote behavioral weight loss randomized clinical trial for type 2 diabetes prevention. Contemp Clin Trials. 2025 Jan;148:107735. doi: 10.1016/j.cct.2024.107735. Epub 2024 Nov 9. PMID 39522630

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The mLife study was a 52-week parallel group randomized behavioral intervention conducted with two sequential cohorts. Recruitment was implemented through targeted advertisements on social media platforms (Facebook and Instagram) and ResearchMatch, directing prospective participants to a study website for eligibility screening. Eligible individuals completed a phone screener and attended a virtual orientation to review procedures and provide informed consent. Recruitment occurred Feb 18-May 20,
Pre-assignment Details: Eligible and interested participants were offered a choice of orientation session times. During the session, the study coordinator provided a comprehensive overview of the study, addressed participant questions, and obtained informed consent. Participants were guided in establishing Fitbit accounts, synchronizing physical activity and weight trackers, and completing baseline assessments. Those who successfully completed baseline procedures were subsequently randomized.
Period: Overall Study
Arm/Group | Gamified mLIFE App Group | Standard mLIFE App
Started | 121 | 122
Completed | 90 | 74
Not Completed | 31 | 48
Not completed — Lost to Follow-up | 23 | 36
Not completed — Withdrawal by Subject | 7 | 12
Not completed — Removed from analysis | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gamified mLIFE App Group | Standard mLIFE App | Total
Number analyzed (Participants) | 121 | 122 | 243
Age, Continuous [Mean (Standard Deviation); unit: years] — Participant's age at baseline assessment Population: Age at baseline assessment
  years | 47.0 (1.0) | 46.4 (1.0) | 46.7 (1.0)
Sex: Female, Male [Count of Participants; unit: Participants] — Sex at baseline assessment
  Participants
    Female | 107 | 112 | 219
    Male | 14 | 10 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 11 | 22
  Not Hispanic or Latino | 110 | 110 | 220
  Unknown or Not Reported | 0 | 1 | 1
Body weight, [Mean (Standard Deviation); unit: kg] — body weight was assessed via the provided Fitbit Aria Air scale (Google)
  kg | 106.8 (2.4) | 104.4 (2.4) | 105.6 (2.4)
Energy intake [Mean (Standard Deviation); unit: kcal/d] — kcals consumed in a day - 24h dietary recall
  kcal/d | 2136.24 (79.64) | 2073.91 (80.1) | 2105.08 (79.9)
Physical Activity [Mean (Standard Deviation); unit: minutes/wk] — Estimated min/wk of moderate-to-vigorous physical activity (MVPA). Fitbit Physical Activity data
  minutes/wk | 261.12 (45.1) | 220.27 (43.19) | 238.0 (44.1)

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Weight
Description: Difference in body weight between follow-up and baseline (follow-up - baseline); positive values indicate weight gain.
Time Frame: 12 months
Population: Intent-to-treat (ITT) analysis was conducted; primary and secondary outcomes were addressed using repeated measure. All participants were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Kg
Arm/Group | Gamified mLIFE App Group | Standard mLIFE App
Number analyzed (Participants) | 121 | 122
Kg | -5.3 (0.64) | -3.49 (0.72)
Statistical Analysis 1: Comparison: Gamified mLIFE App Group vs Standard mLIFE App; Test type: Superiority; p = 0.09, Mixed Models Analysis; Intent-to-treat (ITT) analysis was conducted; primary and secondary outcomes were addressed using repeated measure. Models: time, group, group x time; Mean Difference (Final Values) = -1.81, 95% CI 2-sided [-3.71 to 0.09], Standard Error of Mean 0.97; Intent-to-treat (ITT) analysis was conducted; primary and secondary outcomes were addressed using repeated measure. Models: time, group, group x time

2. Secondary Outcome: Change in Energy Intake
Description: Difference in total energy intake between follow-up and baseline (follow-up - baseline); positive values indicate increased intake.
Time Frame: 12 months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Kcals
Arm/Group | Gamified mLIFE App Group | Standard mLIFE App
Number analyzed (Participants) | 121 | 122
Kcals | -347.73 (91.15) | -257.42 (92.93)

3. Secondary Outcome: Change in Weekly Moderate to Vigorous Physical Activity (MVPA)
Description: Difference in average weekly minutes of moderate-to-vigorous physical activity (MVPA) between follow-up and baseline (follow-up - baseline), derived from Fitbit physical activity data; positive values indicate increased MVPA.
Time Frame: 12 months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: min/wk
Arm/Group | Gamified mLIFE App Group | Standard mLIFE App
Number analyzed (Participants) | 121 | 122
min/wk | -4.66 (23.45) | -3.5 (24.91)

ADVERSE EVENTS:
Time Frame: From enrollment until end of study, up to 52 weeks.
Arm/Group | Gamified mLIFE App Group | Standard mLIFE App
All-Cause Mortality (participants affected / at risk) | 0/121 | 0/122
Serious Adverse Events (participants affected / at risk) | 1/121 | 0/122
Other Adverse Events (participants affected / at risk) | 0/121 | 0/122
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gamified mLIFE App Group (N=121) | Standard mLIFE App (N=122)
Neck injury due to fall (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Fall with neck injury; serious (disability, surgery 12/21/23); not related to intervention; pre-existing spinal disease; withdrew.

LIMITATIONS AND CAVEATS:
The study sample lacked diversity in race/ethnicity and education. Participant attrition was higher than anticipated. Not all potential social support factors were assessed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-07-24): https://cdn.clinicaltrials.gov/large-docs/47/NCT05176847/Prot_SAP_000.pdf
  • Informed Consent Form (2022-01-18): https://cdn.clinicaltrials.gov/large-docs/47/NCT05176847/ICF_001.pdf